CLINICAL TRIAL: NCT00935376
Title: A Pilot Study of Three Short-term Intervention Programs for Sleep Management in Cancer Survivors
Brief Title: Sleep Management in Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Yoshio Nakamura, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 33669; 5R21AT002209 (NIH)
Record Dates: First submitted 2009-06-18; First posted 2009-07-09 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Insomnia
Keywords: Sleep Management; Awareness Training Programs; Mindfulness Meditation; Mind Body Bridging
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Matrix Metalloproteinases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mind-Body Bridging Program (Experimental): The Mind-Body Bridging Program (MBBP) is an awareness training program (ATP)to help individuals improve their health condition and attain a state of well-being. Bridging is the primary technique that facilitates the healing process, by bringing one back to the present moment to experience thoughts, emotions and physical sensations. Bridging aims to reduce the impact of negative thought patterns that contribute to stress in the body.
  Interventions: Behavioral: Mind-Body Bridging Program
- Mindfulness Meditation Program (Experimental): Mindfulness Meditation Program (MMP) is based on Mindfulness-Based Stress Reduction (MBSR), which teaches participants mindfulness skills such as meditation and yoga. Mindfulness may be defined as paying attention in a particular way, on purpose, in the present moment, and nonjudgmentally. The goal of MBSR is to provide participants with experiential tools and mindfulness practices to assist them to become more mindful of themselves, others and their external environment. The techniques are easy to learn and teach individuals to be aware of the present moment, with an open mind in which they can perceive their thoughts, physical sensations, and emotions nonjudgmentally.
  Interventions: Behavioral: Mindfulness Meditation Program
- Sleep Education Program (Active Comparator): The Sleep Education Program (SEP) will serve as the control intervention in which participants will receive classes informing them how to change their habits to improve their sleep, and what to do if they have concerns about their sleep quality.
  Interventions: Behavioral: Sleep Education Program

INTERVENTIONS:
Behavioral: Sleep Education Program — Treatment as usual.
  Other Names: SEP
  Arms: Sleep Education Program
Behavioral: Mind-Body Bridging Program — Bridging aims to reduce the impact of negative thought patterns that contribute to stress in the body.
  Other Names: MBBP
  Arms: Mind-Body Bridging Program
Behavioral: Mindfulness Meditation Program — Mindfulness Meditation Program is based on Mindfulness-Based Stress Reduction, which teaches participants awareness and mindfulness skills using techniques that include a basic meditation practice and yoga.
  Other Names: MMP
  Arms: Mindfulness Meditation Program

SUMMARY:
The pilot project will investigate three short-term intervention programs for sleep management in cancer survivors in a randomized controlled clinical study. Three programs to be examined in the study are:

1. the mind-body bridging program (MBBP),
2. mindfulness meditation program (MMP), and
3. sleep education program (SEP).

DETAILED DESCRIPTION:
This pilot randomized study investigates whether the two awareness training programs (ATP), MBBP and MMP are effective in improving sleep disturbance and in reducing stress in post-treatment cancer patients. The two experimental conditions and the SEP control will each comprise 3 sessions of 2 hr. duration and conducted over 3 consecutive weeks (Week 1-3).

ELIGIBILITY:
Inclusion Criteria:

1. Selection of subjects will be based on their exhibiting sleep disturbance as assessed by a validated sleep questionnaire (MOS Sleep Scale, Hayes et al, 2005).
2. Participant is willing to be randomized to any one of the three interventions, will be willing to attend all three classes, complete self-report questionnaires and collect saliva samples, at pre- and post- treatment, weekly intervals and 2-3 months follow-up.
3. Participant must be English speaking and comprehend information presented during the course of study, including the consent form.

Exclusion Criteria:

1. Underlying psychiatric illness, such as severe or untreated psychopathology (e.g. schizophrenia), or cognitive impairments, neurologic disorders, or dementia.
2. Use of psychotropic medication for any of the above, and for any other unspecified condition.
3. Has had previous exposure to MBBP or MBSR/MMP.
4. Incidence of metastatic cancer
5. Currently taking immuno-suppressants and/or corticosteroids.
6. Compromised physical health, in which individual has impaired mobility: unable to carry out movement exercises, cannot lie down on the floor, kneel, get up from the floor to a standing position.
7. Individuals who are considered at the 'end-of-life' stage of their cancer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2009-05; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Medical Outcomes Study-Sleep Scale | Pre-treatment, Week 1, Week 2, Week 3, Post treatment, Follow up
Functional Assessment of Cancer Therapy - General | Pre-treatment, Post treatment, Follow up
Perceived Stress Scale | Pre-treatment, Week 1, Week 2, Week 3, Post treatment, Follow up

SECONDARY OUTCOMES:
Impact of Event Scale | Pre-treatment, Post treatment, Follow up
Center for Epidemiologic Studies Depression Scale | Pre-treatment, Post treatment, Follow up
Positive Affect-Negative Affect | Pre-treatment, Week 1, Week 2, Week 3, Post treatment, Follow up
Five-factor Mindfulness Questionnaire | Pre-treatment, Post treatment, Follow up
Self-Compassion Scale | Pre-treatment, Post treatment, Follow up
Well-Being Index | Pre-treatment, Week 1, Week 2, Week 3, Post treatment, Follow up

CONTACTS AND LOCATIONS:
Overall Officials: Yoshio Nakamura, Ph.D., Principal Investigator — University of Utah
Locations (1):
- Yoshio Nakamura, Ph.D., Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lipschitz DL, Kuhn R, Kinney AY, Donaldson GW, Nakamura Y. Reduction in salivary alpha-amylase levels following a mind-body intervention in cancer survivors--an exploratory study. Psychoneuroendocrinology. 2013 Sep;38(9):1521-31. doi: 10.1016/j.psyneuen.2012.12.021. Epub 2013 Feb 1. PMID 23375640
- [Derived] Nakamura Y, Lipschitz DL, Kuhn R, Kinney AY, Donaldson GW. Investigating efficacy of two brief mind-body intervention programs for managing sleep disturbance in cancer survivors: a pilot randomized controlled trial. J Cancer Surviv. 2013 Jun;7(2):165-82. doi: 10.1007/s11764-012-0252-8. Epub 2013 Jan 22. PMID 23338490